CLINICAL TRIAL: NCT05919576
Title: The Effectiveness of an Intraoral Scanner With Near-infrared Imaging (Transillumination) Technology for the Detection of Proximal Caries
Brief Title: Near Infrared Technology for the Detection of Proximal Caries
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: ozlemkanar
Record Dates: First submitted 2023-04-05; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Caries,Dental
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (4):
- Visual-Tactile method (VTM): In patients who come for treatment and have a prior appointment, an intraoral examination is performed using visual and tactile examination methods. A total of 639 proximal surfaces of 22 patients are examined by investigators using the visual-tactile method.
- Bitewing Radiography (BTW): Bitewing radiographs available in the hospital system of patients who come to their appointment for treatment are examined. A total 639 proximal surface of 22 patient examined by investigators using bitewing radiography.
- Near-infrared imaging Technology (NIRI): A total 639 proximal surface of 22 patient examined by using the NIRI feature of an intraoral scanner. Patients who came for restorative treatment were asked whether they volunteered in our study. An informed consent form was signed, and then lower and upper jaw scans were made by investigators.
  Interventions: Device: Near infrared imaging
- Panoramic radiography (PR): Panoramic radiographs available in the hospital system of patients who come to their appointment for treatment are examined. A total 639 proximal surface of 22 patient examined by using panoramic radiography.

INTERVENTIONS:
Device: Near infrared imaging — In the study, all volunteers are recorded with the itero Element 5D by activating the NIRI mode. The recording method does not involve ionizing radiation. 850 nm wavelength beams are used.
  Groups: Near-infrared imaging Technology (NIRI)

SUMMARY:
This study aims to determine the effectiveness of an intraoral scanner with near-infrared imaging (NIRI) for the diagnosis of proximal caries.

DETAILED DESCRIPTION:
A total of 639 proximal surfaces (mesial-distal) of 22 volunteers without restoration of premolars and molars were examined. Results were scored for 4 different examination methods; intraoral examination by visual-tactile method (VTM), bitewing radiography (BWR), panoramic radiography (PR) and near-infrared imaging (NIRI). Scoring was made according to the type of lesion (0:no caries, 1:early enamel lesion(EEL), 2:lesion involving the dentin-enamel-junction (DEJ). Data were analyzed with IBM-SPSS-V23. McNemar-Test was used for comparison between the methods. The Kappa Test was used to examine the agreement between two methods in categorical data, and the Fleiss-Kappa Test was used to assess the agreement between more than two methods. The analysis results are presented as frequency(percentage).The significance level was considered p<0.05.

ELIGIBILITY:
Inclusion Criteria

1. Presence of premolar and molar tooth
2. Having an appointment for restorative treatment

Exclusion Criteria

1. Restored proximal surfaces
2. Full mouth crowns and removable dental prothesis

Ages: 14 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients who have treatment appointments at Marmara University Faculty of Dentistry, Department of Restorative Dentistry
Sampling Method: Probability Sample
Enrollment: 639 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-08-29 (Actual)

PRIMARY OUTCOMES:
VTM GROUP (Visual-tactile examination) | 08.08.2022 - 22.08.2022
  Surface codes: Sound surface (0), Enamel lesion (1), Lesions involving DEJ (2). A total of at least 150 surfaces are expected to be examined
Bitewing Radiography | 08.08.2022-22.08.2022
  Surface codes: Sound surface (0), Enamel lesion (1), Lesions involving DEJ (2). A total of at least 150 surfaces are expected to be examined
Panoramic Radiography | 08.08.2022-22.08.2022
  Surface codes: Sound surface (0), Enamel lesion (1), Lesions involving DEJ (2). A total of at least 150 surfaces are expected to be examined
NIRI (Near infrared Imaging Technology) | 08.08.2022-22.08.2022
  Surface codes: Sound surface (0), Enamel lesion (1), Lesions involving DEJ (2). A total of at least 150 surfaces are expected to be examined

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University Faculty of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No